CLINICAL TRIAL: NCT05223231
Title: A Multicenter, Open Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of LBL-019 Monotherapy or Combination Anti-PD-1 Antibody in Patients With Advanced Malignant Tumors
Brief Title: Evaluation of LBL-019 Monotherapy or Combined With Anti-PD-1 Antibody in the Treatment of Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-019-CN001
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-019 (Experimental): singal -arm
  Interventions: Drug: LBL-019 Injection; Drug: anti-PD-1 antibody injection

INTERVENTIONS:
Drug: LBL-019 Injection — initial dose-MTD
  Other Names: LBL-019
Drug: anti-PD-1 antibody injection — provide medicine base on needs
  Other Names: anti-PD-1 antibody

SUMMARY:
This trial is a phase I/II study, which is designed to evaluate the safety, tolerance, pharmacokinetic characteristics, receptor occupancy (RO), immunogenicity and effectiveness of LBL-019 monotherapy or combined with anti-PD-1 antibody in patients with advanced malignant tumors.

DETAILED DESCRIPTION:
This trial is a phase I/II study , which is designed to evaluate the safety, tolerance, pharmacokinetic characteristics, receptor occupancy (RO), immunogenicity and effectiveness of LBL-019 monotherapy or combined with anti-PD-1 antibody in patients with advanced malignant tumors. Approximately 244-486 subjects with advanced malignant tumors will be enrolled.

The study was divided into two phases: Phase I (Part A single therapy dose escalation and Part B combination therapy dose escalation) and Phase II (Part A single therapy dose expansion and Part B combination therapy dose expansion) .

ELIGIBILITY:
Inclusion Criteria:

1.Agree to comply with the trial treatment plan and visit plan, voluntarily agree to sign the informed consent form;

2.18-75 years old (including boundary value), no gender limit;

3. previous standard treatment failed, no standard treatment or standard treatment is not applicable at this stage;

4.The expected survival time is at least 12 weeks;

Exclusion Criteria:

1. Have received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks before using the study drug for the first time；
2. Received any other investigational drug or treatment that is not on the market within 4 weeks prior to the initial use of the investigational drug;
3. Women who are pregnant or breastfeeding;
4. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal. The maximum time is 24 months
  To evaluate the safety, tolerability of LBL-019 monotherapy or combined with anti-PD-1 antibody, which is according to the number of DLT and the number of treatment related AES

SECONDARY OUTCOMES:
Cmax | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal. The maximum time is 24 months
  Maximum serum concentration
immunogenicity | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal. The maximum time is 24 months
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects;
Pharmacodynamics | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal. The maximum time is 24 months
  Receptor occupancy
ORR | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal. The maximum time is 24 months
  Objective Response Rate
DCR | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal. The maximum time is 24 months
  Disease Control Rate
DOR | All subjects signed the informed consent form to the completion of the follow-up period of drug withdrawal. The maximum time is 24 months
  To measure duration of response

CONTACTS AND LOCATIONS:
Overall Officials: caicun zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (6):
- China (6):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Union hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The first affiliated hospital with Nanjing medical university, Nanjing, Jiangsu
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality